CLINICAL TRIAL: NCT00681148
Title: Botulinum Toxin Injection With Prostate Brachytherapy: A Randomized, Placebo-controlled Study Monitoring Urinary Symptoms and PSA
Brief Title: Botulinum Toxin Injection With Prostate Brachytherapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No funding
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Peter T. Nieh, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00009836
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Prostate Cancer; Lower Urinary Tract Symptoms; Radioactive Seed Implantation
Keywords: Prostate specific antigen (PSA); Prostate cancer; Lower urinary tract symptoms; Radioactive seed implantation
MeSH Terms: conditions — Prostatic Neoplasms; Lower Urinary Tract Symptoms | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Botox injection
  Interventions: Drug: Botox injection
- B (Placebo Comparator): Saline injection
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Botox injection — Intraprostatic injection of Botox (100 units for < 30 cc prostate; 200 units for > 30 cc prostate) administering 2 transperineal injections into both lateral lobes of the prostate (25-50 units per injection), just 5-10 mm proximal to the bladder neck.
  Other Names: Botox
  Arms: A
Drug: Saline injection — Saline injection, administering 2 transperineal injections into both lateral lobes of the prostate (1-2 cc per injection), just 5-10 mm proximal to the bladder neck.
  Other Names: NS
  Arms: B

SUMMARY:
The purpose of this study is to see if botox injection into the prostate during seed implantation (brachytherapy) for prostate cancer a) improves urinary symptoms or avoids need for urinary tract instrumentation over the 6-8 month post-operative period when one wants to avoid manipulating the radioactive seeds, and b) speeds up the drop in PSA. Patients will be randomized to botox vs saline injection, at the completion of the seed implantation procedure.

DETAILED DESCRIPTION:
Brachytherapy is a popular treatment modality for localized prostate cancer, where radioactive seeds are implanted through 18 gauge needles into the prostate via a perineal template with rectal ultrasound guidance. The radioactivity is delivered over several months, depending on the isotope used. During this time, there can be exacerbation of urinary voiding symptoms from early edema of the prostate gland due to the implantation procedure, then later from the inflammatory reaction of the radiation. Because the initial acute inflammation may persist for many months despite steadily declining doses of radiation, attempts are made to minimize urinary symptoms prior to brachytherapy with pharmacologic therapy (alpha-blockers) or minimally invasive surgical therapy (transurethral incision or limited transurethral resection to avoid significant distortion of the prostate parenchyma for future seed implantation). Even with these precautions, around 30-40% of brachytherapy patients will still develop voiding symptoms. With such bothersome symptoms, intervention is deferred for at least 8-10 months to avoid distorting the planned field of radiation. Once symptoms develop, various additional pharmacologic measures are employed, such as increased doses of alpha-blockers, medrol steroid taper, and non-steroidal anti-inflammatory agents. Some patients require intermittent self-catheterization or suprapubic catheter for urinary diversion.

Botulinum toxin has been used for cosmetic uses, and has been successfully used for treatment of overactive bladder, external sphincter dyssynergia, and benign prostatic hyperplasia (BPH). The studies with BPH show reduction in symptoms scores, PSA, and prostate volume, the latter from atrophy due to the denervation effect. The response lasts for 6-9 months.

We propose to study botox intraprostatic injection during brachytherapy to see whether this improves urinary symptoms or avoids need for urinary tract instrumentation over this 6-8 month post-operative period when one wants to avoid manipulating the radioactive seeds. We will also monitor PSA, and see if there is any measurable augmentation of PSA decline with botox + Brachytherapy vs Brachytherapy alone. We will randomize patients to botox (100 units for < 30 cc prostate; 200 units for > 30 cc prostate) vs saline injection, administering 2 transperineal injections into both lateral lobes of the prostate (25-50 mg per injection), just 5-10 mm proximal to the bladder neck.

Study design:

N= 60 (30 receive Botox, 30 receive saline)

Followup:

AUA Symptoms scores weekly for 4 weeks, monthly thereafter Medications for urinary symptoms Need for catheterization PSA checked at 1 mo, 3 mo, 6 mo, 9 mo, 1 year, 15 mo, 18 mo, 24 mo

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven prostate cancer undergoing brachytherapy

Exclusion Criteria:

* Prior allergic reaction to botulinum toxin

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Urinary symptoms | Weekly for 4 weeks, monthly thereafter until 1 year

SECONDARY OUTCOMES:
PSA | 1 mo, 3 mo, 6 mo, 9 mo, 1 year, 15 mo, 18 mo, 24 mo

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Nieh, MD, Principal Investigator — Emory University SOM
Locations (1):
- Emory Clinic, Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Background] Lee WR, Hall MC, McQuellon RP, Case LD, McCullough DL. A prospective quality-of-life study in men with clinically localized prostate carcinoma treated with radical prostatectomy, external beam radiotherapy, or interstitial brachytherapy. Int J Radiat Oncol Biol Phys. 2001 Nov 1;51(3):614-23. doi: 10.1016/s0360-3016(01)01707-2. PMID 11597800
- [Background] Wallner K, Merrick G, True L, Sutlief S, Cavanagh W, Butler W. 125I versus 103Pd for low-risk prostate cancer: preliminary PSA outcomes from a prospective randomized multicenter trial. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1297-303. doi: 10.1016/s0360-3016(03)01448-2. PMID 14630265
- [Background] Ansiaux R, Baudelet C, Cron GO, Segers J, Dessy C, Martinive P, De Wever J, Verrax J, Wauthier V, Beghein N, Gregoire V, Buc Calderon P, Feron O, Gallez B. Botulinum toxin potentiates cancer radiotherapy and chemotherapy. Clin Cancer Res. 2006 Feb 15;12(4):1276-83. doi: 10.1158/1078-0432.CCR-05-1222. PMID 16489084
- [Background] Chuang YC, Chancellor MB. The application of botulinum toxin in the prostate. J Urol. 2006 Dec;176(6 Pt 1):2375-82. doi: 10.1016/j.juro.2006.07.127. PMID 17085104
- [Background] Chuang YC, Huang CC, Kang HY, Chiang PH, Demiguel F, Yoshimura N, Chancellor MB. Novel action of botulinum toxin on the stromal and epithelial components of the prostate gland. J Urol. 2006 Mar;175(3 Pt 1):1158-63. doi: 10.1016/S0022-5347(05)00318-6. PMID 16469644